CLINICAL TRIAL: NCT03910205
Title: Gingival Crevicular Fluid Tumor Necrosis Factor-alpha and Interleukin-18 Levels in Children With Gingivitis and Type 1 Diabetes Mellitus
Brief Title: Tumor Necrosis Factor-alpha and Interleukin-18 Levels in Children With Gingivitis and Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Other Study IDs: 2019-062
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-07

CONDITIONS: Periodontal Diseases
Keywords: interleukin-18; gingival crevicular fluid; tumor necrosis factor alpha
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 1 diabetes with gingivitis: Children with type 1 diabetes mellitus and gingivitis
  Interventions: Diagnostic Test: ELISA
- Type 1 diabetes with healthy gingiva: Children with type 1 diabetes mellitus and healthy gingiva
  Interventions: Diagnostic Test: ELISA
- Healthy patients with gingivitis: Systemically healthy patients with gingivitis
  Interventions: Diagnostic Test: ELISA
- Healthy patients with healthy gingiva: Systemically healthy patients with healthy gingiva
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Enzim linked immunoabsorbant assay

SUMMARY:
This study aimed to evaluate the levels of interleukin 18 and tumor necrosis factor-alpha (TNF-α) in gingival crevicular fluid (GCF) of children with type 1 diabetes mellitus and gingivitis.

DETAILED DESCRIPTION:
Eighty eight children (44 with type 1 diabetes mellitus and 44 healty; age range 7-14 years) will be recruited for the study. The children will be classified into four subgroups based on their periodontal status; 1) Children with gingivitis and diabetes mellitus (MG, n=22); 2) Children with type 1 diabetes mellitus with healthy periodontium (MH, n=22); 3)Healthy children with gingivitis (HG, n=22); 4) Healthy children with healthy periodontium (HH, n=22). Probing pocket depth (PPD), gingival index (GI) and plaque index (PI) will be recorded. Interleukin-18 and TNF-α will be analyzed in GCF and saliva samples by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as type 1 diabetes mellitus
* Age between 7 and 14 years

Exclusion Criteria:

* Having another systemic problem except type 1 diabetes mellitus
* Children carrying orthodontic appliances

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 88 Children with diabetes mellitus and systemically healty children with and without gingivitis.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Interleukin-18 level | Baseline
  IL-18

SECONDARY OUTCOMES:
Tnf-alpha level | Baseline
  Tnf-Alpha

CONTACTS AND LOCATIONS:
Overall Officials: Sultan KELES, Dr., Principal Investigator — Dr.
Locations (1):
- Sultan KELES, Aydin, Turkey (Türkiye)